CLINICAL TRIAL: NCT01077908
Title: A Phase III Randomised Study to Investigate the Use of Adoptive Cellular Therapy (ACT) in Combination With Conventional Antiviral Drug Therapy for the Treatment of CMV Reactivation Episodes in Patients Following Allogeneic Haematopoietic Stem Cell Transplant
Brief Title: Cytomegalovirus - Immunoprophylactic Adoptive Cellular Therapy Study
Acronym: CMV-IMPACT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cell Medica Ltd (Industry)
Collaborators: Wellcome Trust (Other); EMAS Pharma (Industry); Commitum AB (Industry); BioAnaLab (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CM-2008-01; 08/H0720/15 (Other: REC); 74928896 (Registry Identifier: ISRCTN); NCT01115816 (obsolete NCT alias)
Record Dates: First submitted 2010-02-26; First posted 2010-03-01 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Cytomegalovirus Infection
Keywords: Adoptive cellular therapy; Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACT plus standard therapy (Experimental): Adoptive Cellular Therapy (ACT) prepared using Multimer or Gamma Catch Selection in combination with standard best available antiviral drug therapy
  Interventions: Biological: Adoptive Cellular Therapy; Drug: Best available antiviral drug therapy
- Best available antiviral drug therapy (Active Comparator)
  Interventions: Drug: Best available antiviral drug therapy

INTERVENTIONS:
Biological: Adoptive Cellular Therapy — CMV-specific T-cells, single infusion at 27 days post-HSCT
  Arms: ACT plus standard therapy
Drug: Best available antiviral drug therapy — 1. Intravenous ganciclovir 5mg/kg twice daily
  2. Oral valganciclovir 900mg twice daily
  3. Intravenous foscarnet 90 mg/kg twice daily

SUMMARY:
The purpose of this study is to evaluate the potential clinical benefit of prophylactic cytomegalovirus (CMV)-specific adoptive cellular therapy following T cell depleted allogeneic hematopoietic stem cell transplantation (HSCT) for reducing recurrent CMV reactivation.

DETAILED DESCRIPTION:
As with other herpes viruses, CMV infection is thought to result most frequently from reactivation of latent virus. Transmission of the virus can also occur from donor marrow infusion or from allogeneic red cell, leukocyte or platelet transfusions. In an allogeneic haematopoietic stem cell (bone marrow) transplant patient who is CMV seropositive or receiving a transplant from a donor who is CMV seropositive, CMV frequently reactivates and disease resulting from the progression of infection is a major cause of infectious morbidity and mortality. CMV infection is a consequence both of the immunosuppression these patients receive and may also reflect delayed immune reconstitution in these patients following transplant.

Existing evidence suggests that adoptive cellular therapy can be an effective approach for treating viral reactivation following allo HSCT, with a minimal risk of inducing GVHD. The major advantage to the patient is likely to be avoidance of extended periods of therapy with antiviral medications that have significant associated morbidities, and sometimes require inpatient care. A proof of efficacy in the sibling donor setting would strengthen the case for extending the therapy to the unrelated donor setting, where both potential risks and benefits are greater. From a pharmacoeconomic viewpoint, the avoidance of the costs associated with these treatment episodes could offset the costs of adoptive cellular therapy. A number of issues remain unresolved. These include the relative contributions of transferred CD4+ and CD8+ T cell populations (which may have direct relevance to the best approach for selection), the issue of whether adoptive cellular therapy improves outcomes in a randomised setting, and equally importantly, the issue of whether such immunotherapies can be delivered outside of the setting of a few academic institutions on a multicentre basis.

These considerations emphasise the importance of undertaking a randomised phase III study of prophylactic adoptive cellular therapy for CMV following T cell depleted allogeneic HSCT from a sibling donor (CMV~IMPACT). There are multiple methods for T cell depletion available, and differences between them will likely have an effect on immune reconstitution. In order to avoid this confounding influence the study will be restricted to patients receiving alemtuzumab-containing conditioning protocols.

In summary, this study is a multicentre, prospective, controlled, open-label 3 arm randomized study comparing 'best-available' standard anti-viral monitoring and therapy alone, with 'best available'anti-viral monitoring and therapy plus prophylactic adoptive cellular therapy (ACT) with cells selected by either the Gamma Catch or Multimer Selection techniques. Patients will be randomised to:

A. Standard best available antiviral drug therapy alone B. Immunoprophylactic (Day 27) ACT prepared using Gamma Catch Selection in combination with standard best available antiviral drug therapy C. Immunoprophylactic (Day 27) ACT prepared using Multimer Selection in combination with standard best available antiviral drug therapy

The study will test the hypothesis that CMV-specific ACT based upon a prescribed T-cell dose/kg recipient body weight, can augment the impaired CMV immune function post-transplant and reduce the number of recurrent reactivations in patients following a primary reactivation event (and thereby reduce the requirement for antiviral drug therapy) without causing an increase in GVHD.

Individual groups will be compared for duration of antiviral therapy and number of reactivation episodes, plus GVHD incidence. Similar analyses will be performed for adoptive cellular therapy versus no therapy (i.e. (B+C) versus A)

ELIGIBILITY:
Inclusion Criteria:

* Suitable participants will be selected from patients already scheduled to undergo a T cell depleted sibling donor HSCT. The criteria will include:
* Age 18 years or older
* Negative markers of Infectious Disease screen
* Recipient of allogeneic HSCT (that incorporates T cell depletion with alemtuzumab) who is CMV seropositive with a CMV seropositive sibling donor
* Informed consent from both donor and patient and to be assessed prior to CMV-specific T cell infusion (confirmed prior to product release):
* Donor engraftment (neutrophils > 0.5x109/l)

Exclusion Criteria:

* Pregnant or lactating women
* Co-existing medical problems that would place the patient at significant risk of death due to GVHD or its sequelae
* HIV infection and to be assessed prior to CMV-specific T cell infusion (confirmed prior to product release):
* Active acute GVHD > Grade I
* Concurrent use of systemic corticosteroids
* Organ dysfunction as measured by

  1. creatinine > 200 uM/l
  2. bilirubin > 50 uM/l
  3. ALT > 3x upper limit of normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2008-07; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
CMV reactivations | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Karl S Peggs, Study Chair — University College London Hospitals
Locations (14):
- United Kingdom (14):
  - Birmingham Heartlands Hospital, Birmingham, West Midlands
  - St James's University Hospital, Leeds, West Yorkshire
  - Queen Elizabeth Hospital, Birmingham
  - Bristol Royal Hospital for Children, Bristol
  - Addenbrookes Hospital, Cambridge
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Royal Liverpool Hospital, Liverpool
  - University College Hospital, London
  - Kings College Hospital, London
  - Royal Free Hospital, London
  - Christie Hospital, Manchester
  - Manchester Royal Infirmary, Manchester
  - City Hospital, Nottingham
  - Southampton General Hospital, Southampton